CLINICAL TRIAL: NCT03271125
Title: Intensive Multimodal Training for Persons With Multiple Sclerosis: Random Controlled Trial
Brief Title: Intensive Multimodal Training for Persons With MS
Acronym: Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treadmill MS
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Rehabilitation; Multiple Sclerosis
Keywords: Intervention; Multiple sclerosis; Treadmill; Mobility
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill group (Experimental): Participants in the experimental group received supervised treadmill training
  Interventions: Behavioral: Treadmill
- Resistance group (Active Comparator): Participants in the control group were treated with Resistance exercises.
  Interventions: Behavioral: Resistance

INTERVENTIONS:
Behavioral: Treadmill — Participants in the experimental group received supervised treadmill training, 4-5 sessions per week. The treatment protocol was aimed at improving participants' resistance, walking velocity, balance and cognitive functions during motor and cognitive (dual) tasks. The treadmill training was carried out without body weight support but if needed the participants were attached to a safety harness.
  Arms: Treadmill group
Behavioral: Resistance — Participants in the control group were treated with Resistance exercises, 4-5 sessions per week. The treatment protocol was aimed at improving strength in muscles involved in walking (hip abductors, quadriceps, plantar flexors, dorsal flexors) according to current guidelines from the American College of Sports Medicine (2009). Three sets of 10 repetitions were performed bilaterally with appropriate weights for each exercise
  Arms: Resistance group

SUMMARY:
The aim of this study was to evaluate the safety, feasibility and preliminary effects of a high-intensity rehabilitative multimodal training protocol carried out on treadmill on walking efficacy, mobility, balance, executive function, fatigue and health-related quality of life in a sample of persons with moderate to severe MS deficit of mobility compared to a control group that received a strengthening program of similar intensity.

DETAILED DESCRIPTION:
Persons with multiple sclerosis can have various deficits, affecting many aspects of physical and cognitive functioning often leading to low levels of physical activity in daily life. These include poor endurance, muscle weakness, incoordination and poor balance and cognitive deficits that can all lead to persistent mobility difficulties in daily life.

Given the importance of exercise and physical activity for persons with multiple sclerosis that are already moderately to severely hampered by their locomotor ability and balance, the setting up of intense functional mobility training that targets the main deficits, in adjunction to a clinical rehabilitation usual care and under close supervision, may be a viable way of increasing the level of physiological health and give a basis for the persons to start their own activity pursuit outside of the rehabilitation clinic. Treadmill walking has several benefits for mobility rehabilitation. First, it is a everyday task, walking. Second it lends itself well to a dual task paradigm where other aspects of mobility, such as equilibrium and cognitive factors can be addressed during walking. Third, even persons with severe walking limitations can train walking at various speeds when on treadmill, holding onto handrails and using safety harnesses that minimize the possibility of adverse events during training. Further, the treadmill paradigm lends itself well to training with progressive task difficulty, numerous rhythmic repetitions, and importantly it can include an aerobic component to improve cardiorespiratory fitness. All of which should lead to improved submaximal exercise tolerance and endurance, more functional mobility and consequently increased ability to carry out activities of daily living.

Methods: A consecutive sample of 42 People with Multiple Sclerosis (PwMS) were recruited from the outpatient/inpatient rehabilitation service of the Don Gnocchi Foundation. The study was conducted in accordance with the Declaration of Helsinki and was approved by the ethics committee of the Don Gnocchi Foundation. Subjects signed an informed consent form before the beginning of the study.

The study design was a two arm randomized 2:1 controlled trial (see study flow chart in Figure 1).

The participants were assessed before and after the rehabilitation period by researchers blinded to group assignment.

Participants in both groups received 15- 20 treatments sessions lasting 30 minutes 5 times per week by experienced physical therapists trained for the study. All participants also followed their usual rehabilitation care protocols as planned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to McDonald's criteria (Polman et al. Ann Neurology 2011)
* EDSS score <= 7
* Free from relapses and steroid treatment for at least 1 month)
* Able to stand 30 seconds,
* Able to walk at least 10 meters independently or with a cane
* Able to understand and follow instructions
* Stable neurological conditions and willingness to participate in the study.

Exclusion Criteria:

* Cardiac pacemaker
* Any pre-existing conditions that affected walking function
* diagnosis of depression or psychotic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2015-05-19 (Actual)

PRIMARY OUTCOMES:
Two minute walking test | Two minutes
  The subjects were instructed to walk at their usual speed for 2 minutes while the distance they covered in 2 minutes was recorded in meters.
Timed up and go test | 1 minute
  The Timed Up & Go test (TUG) is a simple functional test that requires a person to stand up, walk 3m, turn back, and sit down again while being timed.

SECONDARY OUTCOMES:
The Frontal Assessment Battery | 10 minutes
  The Frontal Assessment Battery (FAB) is a short cognitive and behavioral six-subtest battery for the bedside screening of a global executive dysfunction.
Ten meter walking test | 2 minutes
  The 10 meters walking test (10MWT) is a test in which the participant is timed while walking 10m at their comfortable speed.
The Berg Balance Scale | 15 minutes
  The Berg Balance Scale (BBS) is a 14-item scale widely used to assess balance disorders in PwMS. BBS provides information about patient's balance-related abilities.
Dynamic Gait Index | 15 minutes
  The Dynamic Gait Index (DGI) measures gait function and dynamic balance. The eight tasks of this scale include walking, walking with head turns, pivoting, walking over objects, walking around objects, and going upstairs.
The Short Form-12 questionnaire (SF-12) | 10 minutes
  The SF12 is comprised of two domains, physical and mental and gives two composite scores that reflect the perceived health of the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi IRCCS, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Due to ethical restrictions set by the Ethics Committee of Fondazione Don Carlo Gnocchi and the presence of identifying patient information, researchers wishing to access raw data for use in future research studies should write to the Corresponding Author that will apply to the Ethics Committee of Fondazione Don Carlo Gnocchi for approval. Additional data